CLINICAL TRIAL: NCT07128810
Title: Effects of Parent Child Interaction Therapy vs Conventional Parent Led Therapy in the Management of Language Disorders in Children With Down Syndrome
Brief Title: Parent Child Interaction Therapy vs Conventional Parent Led Therapy in Down Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 02114 Ishrat
Record Dates: First submitted 2025-06-11; First posted 2025-08-19 (Actual); Last update posted 2025-08-19 (Actual); Status verified 2025-08

CONDITIONS: Language Disorder
Keywords: Parent Child Interaction Therapy (PCIT); Conventional Parent Led Therapy; Down Syndrome; Language Disorder; Language Management
MeSH Terms: conditions — Language Disorders; Down Syndrome

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Parent Child Interaction Therapy (Experimental)
  Interventions: Other: Parent Child Interaction Therapy
- Conventional Parent Led Therapy (Active Comparator)
  Interventions: Other: Conventional Parent Led Therapy

INTERVENTIONS:
Other: Parent Child Interaction Therapy — Parent was trained in a structured way during two phases of PCIT that are Phase 1: Child Directed Intervention and Phase 2: Parent Directed Intervention to encourage Language Development with frequency of sessions as 12 sessions; minimum 30 mins each day, 3x per week.
  Arms: Parent Child Interaction Therapy
Other: Conventional Parent Led Therapy — Parent was trained in an unstructured way by using different language development strategies (Imitation, Focused Stimulations, Milieu Teaching, and others) to encourage Language Development with frequency of session as 12 sessions; minimum 30 mins each day, 3x per week.
  Arms: Conventional Parent Led Therapy

SUMMARY:
To determine the effect of Parent child interaction therapy vs Conventional Parent Led Therapy in the management of language disorders in Children with Down Syndrome

DETAILED DESCRIPTION:
The most common type of chromosomal defect is Down syndrome (DS), Incidence for Down syndrome in developed countries is 1 of 700 births, however comparatively there is higher incidence in developing countries like Pakistan as one in every 300 births down syndrome occurs. Children with Down syndrome (DS) are prone to learning disorders, morphological unique features and health problems that can include hematological disorders or cardiac problems. Children with down syndrome have unique facial characteristics which can lead difficulties with the biological development of face due to various inheritance factors.

There are significant language delays that are observed among Down syndrome children that can affect their communication ability. The children with Down syndrome typically have a unique language profile in which they have strength in the receptive vocabulary, but show weakness in their expressive language and depth of word knowledge. These children often tend to have more challenges in phonology, morphology, and syntax, whereas the use of language that includes pragmatics are less impaired, but they are still weaker comparatively to the typical developing children.

Children with Down syndrome commonly experience language disorders that affect both expressive and receptive abilities. The language management is essential in the early intervention of Children with Down Syndrome that focuses on many factors, including language therapy that enhances vocabulary and expression. engaging parents as it is vital in order to educate them and provide supportive techniques that can lead to better outcomes.

There are Two prominent interventions for language problems are Parent-Child Interaction Therapy (PCIT) and Clinician-Directed Therapy (CDT). The main focus of PCIT is to enhance the quality of the parent-child relationship and improving behavioral interactions through structured coaching. The aim of this method to create a more supportive and engaging environment for the child's language development. Where as comparatively CDT is direct therapist-led sessions that are designed to target specific language skills based on structured activities and exercises.

PCIT is structured, behavior-change intervention for young children between the ages of 2 and 7 years helping parents adopt less directive, positively engaging approaches that may improve parent-reported child communication skills. PCIT includes two stages; the first one is Child-Directed Interaction (CDI) for enhancing positive interactions and reinforcing desired behaviors, while the second stage is based on effective discipline strategies, Parent- Directed Interaction (PDI). From recent evidence it was reported that parent interaction skills and children's language the outcomes are significantly improved in post PCIT cases.

The Child-Directed Interaction (CDI) phase of Parent-Child Interaction Therapy focuses on building positive relationships, mainly for children with delayed language development. In this phase, parents engage in child-led play, using PRIDE skills like reflecting their child's phrases and providing descriptive language to positively enhance communication and reduce control. The Parent-Directed Interaction phase then shifts to teaching parents effective behavior management strategies. This includes setting clear expectations, using consistent discipline, and applying tools like timeouts and positive reinforcement.

Parents practice these techniques during therapy sessions, receiving feedback through video analysis, which helps them refine their approach and build confidence. As the interactions become more complex, the therapist's support gradually lessens, allowing parents to independently apply what they've learned.

In contrast conventional parent-mediated therapy is done in unstructured environment in which parents are active agents in the therapeutic strategies to enhance their child's communications and social skills. This approach equips parents with the competency to facilitate learning during daily interactions, which in turn helps the child achieve better developmental outcomes.

This parent-mediated therapy efficiently trains parents to make use of techniques that will contribute to the development of impaired children's language. Research has shown the influence of this strategy on receptive and expressive language, implying that a long-lasting effect can be accounted for in these studies of such interventions over some time.

Comparing the effects of Parent-Child Interaction Therapy with conventional parent-led therapy for managing language disorders in children with Down Syndrome will help optimize the intervention strategies. PCIT is more systematic and evidence-based, focusing on enhancing parent-child interactions through specific phases that have been shown to improve communication skills and behavioral outcomes. Conventional parent-led therapies provide flexible, individualized techniques for vocabulary and sentence structure building through daily interactions. The two methods are compared to determine which one will more effectively support language development, taking into account the structured framework of PCIT and the adaptability of traditional therapies. This comparison is crucial for clinical practice and will help guide families in selecting the intervention that best meets their child's specific needs.

ELIGIBILITY:
Inclusion Criteria:

* Children with Down Syndrome

  * Children diagnosed with Down Syndrome
  * Children that have acquired pre linguistic skills like eye contact, non-verbal imitation, joint attention, turn taking
  * Children having nonverbal intentional communication.
  * Children having core receptive vocabulary of 50 words.
* Parents

  * Mother or father of a child with Down syndrome.

Exclusion Criteria:

- Children with Down Syndrome

* Children with co morbid conditions like hearing and visual impairment.
* Child concurrently enrolled in other Speech therapy programs. Parents
* Parents previously trained for PCIT.

Ages: 1 Year to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 16 (Actual)
Dates: Start 2025-03-15 (Actual); Primary Completion 2025-05-29 (Actual); Study Completion 2025-05-30 (Actual)

PRIMARY OUTCOMES:
MacArthur-Bates Communicative Development Inventories (CDI) - Semantics composite | 1st session, 6th session and 12th session (The Duration of each session is 45 minutes)
  The MacArthur-Bates Communicative Development Inventories (CDI) is a standardized, parent-report tool used to assess early sementic development in children. It consist of two sections: word comprehension and word production.
  At the baseline (1st session), this tool is administered to establish the child's initial vocabulary level.
  At the midpoint (6th session), scores are calculated based on the number of words the child understands and produces, allowing for measurement of progress.
  At the end of the intervention (12th session), the CDI is administered again to evaluate changes in vocabulary comprehension and production.
  The Duration of each session was 45mins This tool provides a reliable means of tracking language acquisition and measuring the effectiveness of the intervention over time.

CONTACTS AND LOCATIONS:
Overall Officials: Soabah Wasim, MS SLP, Principal Investigator — Riphah International University
Locations (1):
- Riphah International University Gulberg Green, Islamabad, Federal, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cronin SM. An effectiveness study of a parent-child interaction therapy with children with Down syndrome.
- [Background] Roberts MY, Curtis PR, Sone BJ, Hampton LH. Association of Parent Training With Child Language Development: A Systematic Review and Meta-analysis. JAMA Pediatr. 2019 Jul 1;173(7):671-680. doi: 10.1001/jamapediatrics.2019.1197. PMID 31107508
- [Background] Agarwal Gupta N, Kabra M. Diagnosis and management of Down syndrome. Indian J Pediatr. 2014 Jun;81(6):560-7. doi: 10.1007/s12098-013-1249-7. Epub 2013 Oct 15. PMID 24127006
- [Background] Spellun A, Harstad E, Hojlo M, Milliken A, Pawlowski K, Sideridis G, Baumer N. Cross-Sectional Analysis of Caregiver-Reported Expressive Language Profiles and Associated Covariates in Individuals with Down Syndrome. J Dev Behav Pediatr. 2024 Jan 1;45(1):e63-e71. doi: 10.1097/DBP.0000000000001236. Epub 2023 Dec 20. PMID 38117678
- [Background] Bittles AH, Bower C, Hussain R, Glasson EJ. The four ages of Down syndrome. Eur J Public Health. 2007 Apr;17(2):221-5. doi: 10.1093/eurpub/ckl103. Epub 2006 Jul 19. PMID 16857692
- [Background] Yamauchi Y, Aoki S, Koike J, Hanzawa N, Hashimoto K. Motor and cognitive development of children with Down syndrome: The effect of acquisition of walking skills on their cognitive and language abilities. Brain Dev. 2019 Apr;41(4):320-326. doi: 10.1016/j.braindev.2018.11.008. Epub 2018 Nov 28. PMID 30503574